CLINICAL TRIAL: NCT03182985
Title: The Impact of Time Restricted Feeding (TRF) in Improving the Health of Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, Pam Taub, MD, Associate Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UCSD IRB 170504
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Weight Loss; Metabolic Syndrome; Overweight and Obesity
MeSH Terms: conditions — Weight Loss; Metabolic Syndrome; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Time Restricted Feeding (Experimental): Patients will reduce daily oral intake to 10 hours per day
  Interventions: Behavioral: Time Restricted Feeding

INTERVENTIONS:
Behavioral: Time Restricted Feeding — Participants will reduce the amount of time they eat to 10 hours per day and will log their dietary intake using a smartphone application.

SUMMARY:
The investigators intend to measure the health impact of a dietary intervention known as time restricted feeding (TRF) on patients with metabolic syndrome (three or more of: increased waist circumference, abnormal cholesterol levels, elevated blood pressure, or elevated blood sugar). The investigators will enroll patients with metabolic syndrome who eat for ≥ 14 hours per day and will ask participants to reduce daily oral intake to 10 hours per day. The investigators will assess the impact of this dietary change using measures obtained before and after a 12 week intervention period, including body mass index, blood pressure, various lab parameters and blood sugar levels (assessed using a continuous glucose monitor). The investigators will assess for compliance with TRF using a Smart Phone application (myCircadianClock (mCC) app).

ELIGIBILITY:
Inclusion Criteria:

1. Waist circumference ≥ 102 cm (Men) or ≥ 88 cm (Women).
2. Triglycerides ≥ 150 mg/dL (or on drug treatment for elevated triglycerides).
3. Reduced HDL-C < 40 mg/dL (Men), < 50 mg/dL (Women) (or on drug treatment for reduced HDL-C).
4. Elevated blood pressure, systolic blood pressure ≥ 130 mmHg and/or diastolic blood pressure ≥ 85 mmHg (or treatment with antihypertensive drug with history of hypertension).
5. Elevated fasting glucose ≥ 100 mg/dL (or drug treatment of elevated blood glucose).
6. Age ≥18 years.
7. If patients are on cardiovascular medications (HMG coenzyme A reductase inhibitors (statins), other lipid modifying drugs (including over the counter drugs such as red yeast rice and fish oil), anti-hypertensive, anti-diabetes drugs), no dose adjustments will be allowed during the study period
8. Own a Smartphone with Apple iOperating System (OS) or Android OS. Baseline eating period is ≥ 14 hours per day.

Exclusion Criteria:

1. Pregnant or breast-feeding.
2. Caregiver for a dependent requiring frequent nocturnal care/sleep interruptions. Shift workers with variable (e.g. nocturnal) hours.
3. Planned international travel during the study period.
4. Active tobacco abuse or history of treatment for alcohol abuse,
5. Known inflammatory and/or rheumatologic disease,
6. Known history of familial hypercholesterolemia,
7. History of major adverse cardiovascular event within the past 1 year (acute coronary syndrome (ACS), percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack (TIA))
8. Uncontrolled arrhythmia (i.e. rate-controlled atrial fibrillation/atrial flutter are not exclusion criteria)
9. History of sudden cardiac death (SCD) or implantable cardiac defibrillator (ICD) implantation for any reason,
10. Known history of thyroid or adrenal disease,
11. Any history of malignancy,
12. Known history of type I diabetes,
13. Known history of major immune disease,
14. Eating disorder or bile syndrome,
15. History of cirrhosis
16. History of stage 4 or 5 chronic kidney disease or requiring dialysis
17. History of chronic obstructive pulmonary disease (COPD)
18. Known active infectious diseases,
19. Currently enrolled in a weight-loss or weight-management program,
20. On a special or prescribed diet for other reasons (e.g. Celiac disease),
21. Currently taking any medication that is meant for, or has known effect on, appetite,
22. Any history of surgical intervention for weight management,
23. History of venous thromboembolism.
24. Uncontrolled psychiatric disorder (including history of hospitalization for psychiatric illness)
25. History of known clotting or bleeding disorder(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Mean blood glucose | 12 weeks
  Measured using a continuous glucose monitoring (CGM) device

SECONDARY OUTCOMES:
Insulin, triglycerides, hs-CRP levels | 12 weeks
  Measured by blood test

CONTACTS AND LOCATIONS:
Overall Officials: Pam Taub, MD, Principal Investigator — UCSD
Locations (1):
- UCSD, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaix A, Zarrinpar A, Miu P, Panda S. Time-restricted feeding is a preventative and therapeutic intervention against diverse nutritional challenges. Cell Metab. 2014 Dec 2;20(6):991-1005. doi: 10.1016/j.cmet.2014.11.001. PMID 25470547
- [Background] Gill S, Le HD, Melkani GC, Panda S. Time-restricted feeding attenuates age-related cardiac decline in Drosophila. Science. 2015 Mar 13;347(6227):1265-9. doi: 10.1126/science.1256682. PMID 25766238